CLINICAL TRIAL: NCT06176573
Title: Pre-operative Versus Post-operative Vaginal Cleansing With Chlorhexidine Solution in Prevention of Post-Cesarean Section Infectious Morbidity at a Teaching Hospital in a Resource Poor Setting: A Randomized Trial.
Brief Title: Pre-operative Versus Post-operative Vaginal Cleansing With Chlorhexidine Solution in Prevention Post-Cesarean Section Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Nwali Matthew Igwe, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PVPVC2023CT
Record Dates: First submitted 2023-12-08; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Post Cesarean Infectious Morbidity
MeSH Terms: interventions — Chlorhexidine; Antibiotic Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First arm - Pre-operative vaginal cleansing with chlorhexidine (Active Comparator): Had vaginal cleansing with chlorhexidine prior to cesarean section and were monitored for infectious morbidity.
  Interventions: Procedure: Chlorhexidine
- Second arm - Post-operative vaginal cleansing with chlorhexidine (Active Comparator): Had vaginal cleansing with chlorhexidine after cesarean section and were monitored for infectious morbidity.
  Interventions: Procedure: Chlorhexidine

INTERVENTIONS:
Procedure: Chlorhexidine — Pre-operative and post-operative vaginal cleansing.
  Other Names: Antibiotic prophylaxis

SUMMARY:
Maternal infectious morbidity is a common complication of cesarean delivery, especially in a poor recourse setting like ours. This study was done to compare the effectiveness of preoperative vaginal cleansing with immediate postoperative vaginal cleansing with chlorhexidine solution in preventing post-cesarean infectious morbidities. Randomized trial involving 120 consented women who had elective or emergency cesarean sections at term, 60 in each group. Group 1 had preoperative while group 2 had postoperative vaginal cleansing with 1% chlorhexidine.

DETAILED DESCRIPTION:
Background: Maternal infectious morbidity is a common complication of cesarean delivery, especially in a poor recourse setting like ours. This study was done in a tertiary hospital in Abakaliki, Ebonyi State, Southeast Nigeria over a period of 5 months. The State is inhabited mainly by rural farmers and petty traders. Literacy is low and poverty is common with poor maternal health indices.

Aim: To compare the effectiveness of preoperative vaginal cleansing with immediate postoperative vaginal cleansing with chlorhexidine solution in preventing post-cesarean infectious morbidities.

Method: Randomized trial involving 120 consented women who had elective or emergency cesarean sections at term, 60 in each group. Group 1 had preoperative while group 2 had postoperative vaginal cleansing with 1% chlorhexidine. Research Randomizer software was used to generate 120 numbers. Sixty numbers were randomly generated from a pool of 120 numbers and were assigned to group 1 while the remaining 60 numbers were automatically assigned to group 2. Both groups received antibiotics and anterior abdominal wall scrubbing. There were monitored for symptoms and signs of endometritis, wound infection and pyrexia till discharge.

ELIGIBILITY:
Inclusion Criteria:

* Those that gave consent
* Term pregnancy

Exclusion Criteria:

* Refusal of consent
* Antepartum hemorrhage
* Cord prolapse
* Fetal distress
* Anemia in pregnancy
* Presence of fever and chorioamnionitis

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
infectious morbidity | six (6) weeks.
  development of infectious morbidity following cesarean section after vaginal cleansing.

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria